CLINICAL TRIAL: NCT07184242
Title: Multi-joint Strength Exercises and Proprioceptive Somatosensory Stimulation on Pain, Function, Quality of Life, Sleep Quality, and Psychosocial Factors in Patients Over 60 Years of Age With Chronic Rotator Cuff-related Shoulder Pain
Brief Title: Strength Training and Proprioceptive Stimulation on Pain, Function, Quality of Life, Sleep Quality, and Psychosocial Factors in Older Adults With Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UUJA
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): A control group (CG) will be evaluated in the pre- and post-study phases. Participants assigned to this group will continue their usual conventional treatment in the rehabilitation service to which they are assigned. They will also receive general advice on the positive effects of regular physical activity on their therapeutic process, based on the World Health Organization guidelines for those over 60 years of age.
- Experimental Group (Experimental): The experimental group will participate in a 12-week therapeutic exercise program designed to complement conventional treatment. Following an initial evaluation and informed consent, participants will attend two supervised group sessions per week, each lasting 50-60 minutes. These sessions will combine proprioceptive somatosensory exercises, multi-joint strength training, and specific complementary movements. Exercise loads will be carefully individualized, taking into account each participant's pain threshold, physical characteristics, clinical stage, and symptoms. A structured progression will be ensured by applying progressive overload through systematic changes in repetitions, external resistance, and range of motion. To reinforce the supervised training, participants will also carry out two to three additional home sessions per week, supported with educational materials, a personal logbook, and an adherence diary to encourage continuity and engagement throughout the intervention.
  Interventions: Other: Shoulder Exercise & Proprioceptive Training Program

INTERVENTIONS:
Other: Shoulder Exercise & Proprioceptive Training Program — The study includes two intervention modalities. The experimental group will combine conventional treatment with a structured 12-week therapeutic exercise program, with two supervised group sessions per week (50-60 minutes), which will include proprioceptive somatosensory work, multi-joint strength exercises, and adapted specific movements. Progression will be individually adjusted based on each participant's pain tolerance, physical condition, and clinical progress, complemented by home activities and supporting educational materials.
  The control group will receive only conventional treatment provided at their rehabilitation center and general guidelines on the benefits of physical activity according to WHO recommendations for people over 60 years of age.
  Arms: Experimental Group

SUMMARY:
A single-blind randomized clinical trial with a pretest posttest design is proposed in adults over 60 years of age with chronic shoulder pain due to rotator cuff involvement. Participants will be divided into an experimental group that will receive a multi-joint strength exercise program along with proprioceptive somatosensory stimulation plus conventional treatment for 12 weeks and a control group that will only receive conventional treatment. Assessments will be performed at the beginning and end of the intervention by measuring pain with the NPRS and BPI SF scales, psychosocial factors with PCS FABQ PVAQ and TSK 11, functional disability with the Shoulder Rating Questionnaire, sleep quality with the Pittsburgh Index, and physical function with the Back Scratch Test, goniometry and inclinometer, shoulder dynamometry, and manual grip. It is expected that the combined intervention will significantly improve pain, associated psychosocial factors, quality of life, sleep, and functional capacity of participants.

ELIGIBILITY:
Inclusion Criteria:

* People over 60 years of age.
* Be able to understand the instructions and answer the questionnaires designed for this study, as well as participate in the established physical tests.
* People with rotator cuff-related shoulder pain (RCSRP) of at least 3 months' duration.
* Sign informed consent to participate in the study.
* Possible medical diagnoses to categorize you as RCSRP:
* Subacromial syndrome or subacromial pain syndrome.
* Subacromial impingement.
* Rotator cuff tendinopathy/tendinitis/tendinosis.
* Subdeltoid/subacromial bursitis.
* Non-traumatic partial tears of a rotator cuff tendon affecting less than 50% of the tendon thickness.
* Mild/moderate intrasubstance rotator cuff tears.

Exclusion Criteria:

* Complete/massive rotator cuff tears.
* Corticosteroid injections within the last 6 weeks.
* Recent surgery on that shoulder or planned surgery within the next 3 months.
* Bilateral shoulder pain.
* Presence of glenohumeral fractures or osteoarthritis confirmed by radiographic examination.
* Psychiatric illnesses or central or peripheral neurological disorders that make it difficult to grasp, cooperate, or follow instructions during the procedure.
* Individuals with an absolute contraindication to moderate-to-high-intensity physical exercise based on prior medical testing.
* Presence of severe difficulties with gait, balance, or functional activity, or hearing or vestibular disorders that prevent the performance of the prescribed exercises.
* Visual disturbances that cannot be corrected with glasses, contact lenses, or surgery.
* Being enrolled in another physical exercise or treatment program during the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | Up to twelve weeks
  The NPRS is an 11-point numeric scale (0-10) used to assess pain intensity. Participants indicate their current level of pain, with 0 representing "no pain" and 10 representing "worst imaginable pain." It will be applied to capture the sensory-discriminative dimension of pain.
Brief Pain Inventory - Short Form (BPI-SF) | Up to twelve weeks
  The BPI-SF is a self-administered questionnaire that evaluates pain severity and pain interference with daily activities. It complements the NPRS by covering affective and functional dimensions of the pain experience.
Algometry (Pressure Pain Thresholds) | Up to twelve weeks
  Pressure algometry will be used to determine pain thresholds to pressure stimuli. It allows the quantification of mechanical sensitivity and the evaluation of changes in pain perception.
Pain Catastrophizing Scale (PCS) | Up to twelve weeks
  The PCS is a validated questionnaire that measures catastrophic thinking related to pain through three subscales: rumination, magnification, and helplessness. Higher scores indicate greater pain catastrophizing.
Fear-Avoidance Beliefs Questionnaire (FABQ) | Up to twelve weeks
  The FABQ evaluates fear-avoidance beliefs regarding physical activity and work. It identifies how fear of pain may influence behavior and functional limitations.
Pain Vigilance and Awareness Questionnaire (PVAQ-9) | Up to twelve weeks
  The PVAQ-9 assesses hypervigilance and attentional focus on pain sensations. It quantifies the degree to which individuals monitor, detect, and are alert to pain-related stimuli.
Tampa Scale for Kinesiophobia (TSK-11) | Up to twelve weeks
  The TSK-11 short version is a self-reported questionnaire measuring kinesiophobia, i.e., the fear of movement due to pain or risk of injury. It captures cognitive and emotional aspects of avoidance behavior.
Shoulder Rating Questionnaire (SRQ) | Up to twelve weeks
  The SRQ is a disease-specific tool validated in Spanish that measures functional disability related to shoulder pain. It evaluates domains such as pain, daily activity limitations, and overall shoulder function.
Pittsburgh Sleep Quality Index (PSQI) | Up to twelve weeks
  The PSQI is a widely used questionnaire to assess sleep quality over the previous month. It includes seven components (subjective sleep quality, latency, duration, efficiency, disturbances, medication use, and daytime dysfunction), providing a global score of sleep quality.
Back Scratch Test | Up to twelve weeks
  The Back Scratch Test evaluates shoulder flexibility and range of motion by measuring the distance between the hands behind the back. It is a simple field test for functional shoulder mobility.
Goniometry (Shoulder Range of Motion) | Up to twelve weeks
  A goniometer will be used to measure active range of motion in flexion, abduction, and rotations of the shoulder. The inclinometer option will ensure precise angular assessment.
Handheld Dynamometry | Up to twelve weeks
  Isometric muscle strength of the main shoulder movements (flexion, abduction, rotation) and handgrip strength will be measured with a handheld dynamometer, providing objective data on functional capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- ICOT rehabilitation centers, Las Palmas de Gran Canaria, Spain